CLINICAL TRIAL: NCT04500873
Title: Diagnostic Performance of a Recombinant Polymerase Amplification Test - Lateral Flow (RPA-LF) for Cutaneous Leishmaniasis in an Endemic Setting of Colombia
Brief Title: Performance of RPA-LF for Cutaneous Leishmaniasis
Acronym: RPA-LF
Status: Completed | Type: Observational
Sponsor: Centro Internacional de Entrenamiento e Investigaciones Médicas (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 222972553501; 222972553501 (Other: COLCIENCIAS)
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cutaneous Leishmaniasis (Diagnosis)
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CL is public health in the Americas, diagnostic confirmation is required to start treatment, however current diagnostic methods have several limitations and its access is limited.

Technical requirements of conventional molecular diagnostics and costs preclude their routine use in primary care facilities in rural areas. A recently developed method of Isothermal Recombinase Polymerase Amplification (RPA) targeting Leishmania kinetoplast DNA, has shown high accuracy in detecting Leishmania Viannia spp. We evaluated the diagnostic performance of the RPA-LF test in a laboratory reference center and field scenario with community participation.

DETAILED DESCRIPTION:
CL is public health in the Americas with an average of 55,000 cases per year between 2001 - 2018 in 17 countries, which mainly occur in rural areas with an average of 55,000 cases per year between 2001 - 2018 in 17 countries. Diagnostic confirmation is required to start treatment, however current diagnostic methods have several limitations, and sometimes it is necessary to perform confirmatory tests that are not available in endemic areas.

Several molecular diagnostic tests have been developed for the diagnosis of CL, however, the technical requirements and costs of sample processing by conventional or quantitative PCR preclude their routine use in primary care facilities in resource-constrained settings. A recently developed method of Isothermal Recombinase Polymerase Amplification (RPA) targeting Leishmania kinetoplast DNA, coupled with lateral flow (LF) immunochromatographic strip has shown high accuracy in detecting Leishmania Viannia spp. We evaluated the diagnostic performance of RPA-LF test in two scenarios: laboratory reference center and field with community participation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with 2 years of age and over of any ethnic group
* Ulcerated skin lesions compatible with cutaneous leishmaniasis with two or more weeks of duration
* Approval of informed consent

Exclusion Criteria:

* Mucosal leishmaniasis
* Clinical presentations of cutaneous leishmaniasis different of ulcerated lesions

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with cutaneous lesions compatible with cutaneous leishmaniasis from South west of Colombia
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Performance of RPA-LF compared with the composite gold standard (smear, culture, histopathology, and q-PCR-18S) in two scenarios: reference laboratory and field. | Feb 2018 - August 2020
  Sensitivity, specificity, predictive values (positive and negative) and likelihood ratios with their corresponding 95% confidence intervals will be calculated in both scenarios. We define as true positive (TP) when at least one of the gold standard tests (smear, culture, histopathology or q-PCR-18S) and RPA-LF are positive. A patient was considered true negative (TN) when at least smear, q-PCR-18S were negative and, culture and RPA-LF also resulted in negative.
  Reference lab scenario refers to when the samples are obtained by highly trained technicians (auxiliary nurses) in urban areas localized in Tumaco in a Primary Health facility and send to the reference center in Cali to be processed. In Reference center samples are taken and processed by an expert microbiologist.
  Field refers when the samples are obtained by trained community health workers (CHW) and processed by a non-expert field technician in Tumaco in a primary health facility.

SECONDARY OUTCOMES:
Performace of RPA-LF compared with 4 aditional reference standards in both scenarios. | Feb 2018 - August 2020
  Sensitivity, specificity , predictive values (positive and negative) and likelihood ratios and 95% confidence intervals will be also estimated using 4 reference tests 1)the same as the gold standard but without qPCR; 2) lesion smear microscopy and culture; 3) lesion smear microscopy read in reference lab and 4) lesion smear microscopy read in the primary health facility in both scenarios.

CONTACTS AND LOCATIONS:
Locations (1):
- Corporación Centro Internacional de entrenamiento e Investigaciónes Médicas, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alvar J, Velez ID, Bern C, Herrero M, Desjeux P, Cano J, Jannin J, den Boer M; WHO Leishmaniasis Control Team. Leishmaniasis worldwide and global estimates of its incidence. PLoS One. 2012;7(5):e35671. doi: 10.1371/journal.pone.0035671. Epub 2012 May 31. PMID 22693548
- [Background] Reveiz L, Maia-Elkhoury AN, Nicholls RS, Romero GA, Yadon ZE. Interventions for American cutaneous and mucocutaneous leishmaniasis: a systematic review update. PLoS One. 2013 Apr 29;8(4):e61843. doi: 10.1371/journal.pone.0061843. Print 2013. PMID 23637917
- [Background] Gomes CM, Paula NA, Morais OO, Soares KA, Roselino AM, Sampaio RN. Complementary exams in the diagnosis of American tegumentary leishmaniasis. An Bras Dermatol. 2014 Sep-Oct;89(5):701-9. doi: 10.1590/abd1806-4841.20142389. PMID 25184908
- [Background] Weigle KA, de Davalos M, Heredia P, Molineros R, Saravia NG, D'Alessandro A. Diagnosis of cutaneous and mucocutaneous leishmaniasis in Colombia: a comparison of seven methods. Am J Trop Med Hyg. 1987 May;36(3):489-96. doi: 10.4269/ajtmh.1987.36.489. PMID 2437815
- [Background] Boggild AK, Ramos AP, Espinosa D, Valencia BM, Veland N, Miranda-Verastegui C, Arevalo J, Low DE, Llanos-Cuentas A. Clinical and demographic stratification of test performance: a pooled analysis of five laboratory diagnostic methods for American cutaneous leishmaniasis. Am J Trop Med Hyg. 2010 Aug;83(2):345-50. doi: 10.4269/ajtmh.2010.09-0414. PMID 20682880
- [Background] Braz LMA. Tegumentary leishmaniasis diagnosis: what happened with MST (Montenegro Skin Test) in Brazil? Rev Inst Med Trop Sao Paulo. 2019 Mar 11;61:e17. doi: 10.1590/S1678-9946201961017. No abstract available. PMID 30864622
- [Background] Aronson N, Herwaldt BL, Libman M, Pearson R, Lopez-Velez R, Weina P, Carvalho EM, Ephros M, Jeronimo S, Magill A. Diagnosis and Treatment of Leishmaniasis: Clinical Practice Guidelines by the Infectious Diseases Society of America (IDSA) and the American Society of Tropical Medicine and Hygiene (ASTMH). Clin Infect Dis. 2016 Dec 15;63(12):e202-e264. doi: 10.1093/cid/ciw670. Epub 2016 Nov 14. PMID 27941151
- [Background] de Vries HJ, Reedijk SH, Schallig HD. Cutaneous leishmaniasis: recent developments in diagnosis and management. Am J Clin Dermatol. 2015 Apr;16(2):99-109. doi: 10.1007/s40257-015-0114-z. PMID 25687688
- [Background] Adams ER, Gomez MA, Scheske L, Rios R, Marquez R, Cossio A, Albertini A, Schallig H, Saravia NG. Sensitive diagnosis of cutaneous leishmaniasis by lesion swab sampling coupled to qPCR. Parasitology. 2014 Dec;141(14):1891-7. doi: 10.1017/S0031182014001280. Epub 2014 Aug 11. PMID 25111885
- [Background] Motazedian H, Karamian M, Noyes HA, Ardehali S. DNA extraction and amplification of leishmania from archived, Giemsa-stained slides, for the diagnosis of cutaneous Leishmaniasis by PCR. Ann Trop Med Parasitol. 2002 Jan;96(1):31-4. doi: 10.1179/000349802125000484. PMID 11989531
- [Background] Jara M, Adaui V, Valencia BM, Martinez D, Alba M, Castrillon C, Cruz M, Cruz I, Van der Auwera G, Llanos-Cuentas A, Dujardin JC, Arevalo J. Real-time PCR assay for detection and quantification of Leishmania (Viannia) organisms in skin and mucosal lesions: exploratory study of parasite load and clinical parameters. J Clin Microbiol. 2013 Jun;51(6):1826-33. doi: 10.1128/JCM.00208-13. Epub 2013 Apr 3. PMID 23554201
- [Background] Weigle KA, Labrada LA, Lozano C, Santrich C, Barker DC. PCR-based diagnosis of acute and chronic cutaneous leishmaniasis caused by Leishmania (Viannia). J Clin Microbiol. 2002 Feb;40(2):601-6. doi: 10.1128/JCM.40.2.601-606.2002. PMID 11825977
- [Background] Faber WR, Oskam L, van Gool T, Kroon NC, Knegt-Junk KJ, Hofwegen H, van der Wal AC, Kager PA. Value of diagnostic techniques for cutaneous leishmaniasis. J Am Acad Dermatol. 2003 Jul;49(1):70-4. doi: 10.1067/mjd.2003.492. PMID 12833011
- [Background] Bensoussan E, Nasereddin A, Jonas F, Schnur LF, Jaffe CL. Comparison of PCR assays for diagnosis of cutaneous leishmaniasis. J Clin Microbiol. 2006 Apr;44(4):1435-9. doi: 10.1128/JCM.44.4.1435-1439.2006. PMID 16597873
- [Background] Saldarriaga OA, Castellanos-Gonzalez A, Porrozzi R, Baldeviano GC, Lescano AG, de Los Santos MB, Fernandez OL, Saravia NG, Costa E, Melby PC, Travi BL. An Innovative Field-Applicable Molecular Test to Diagnose Cutaneous Leishmania Viannia spp. Infections. PLoS Negl Trop Dis. 2016 Apr 26;10(4):e0004638. doi: 10.1371/journal.pntd.0004638. eCollection 2016 Apr. PMID 27115155
- [Background] Drain PK, Hyle EP, Noubary F, Freedberg KA, Wilson D, Bishai WR, Rodriguez W, Bassett IV. Diagnostic point-of-care tests in resource-limited settings. Lancet Infect Dis. 2014 Mar;14(3):239-49. doi: 10.1016/S1473-3099(13)70250-0. Epub 2013 Dec 10. PMID 24332389
- [Derived] Cossio A, Jojoa J, Castro MDM, Castillo RM, Osorio L, Shelite TR, Gore Saravia N, Melby PC, Travi BL. Diagnostic performance of a Recombinant Polymerase Amplification Test-Lateral Flow (RPA-LF) for cutaneous leishmaniasis in an endemic setting of Colombia. PLoS Negl Trop Dis. 2021 Apr 28;15(4):e0009291. doi: 10.1371/journal.pntd.0009291. eCollection 2021 Apr. PMID 33909619